CLINICAL TRIAL: NCT00114985
Title: A Phase II Study of Late Rectal Toxicity Following 3-D Conformal External Beam Radiation Therapy Performed Using a Prostate Immobilization Device
Brief Title: Prostate Immobilization Device Used During Radiation Treatments to Decrease Rectal Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anthony V. D'Amico, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-050
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Total Androgen Suppression; Simulation; 3-D Conformal External Beam Radiation Therapy; Intra-rectal immobilization device; Quality of Life Assessment Questionnaire; Rectal Bleeding; Late effects
MeSH Terms: conditions — Prostatic Neoplasms; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Prostate Immobilization Device — Device placed during radiation treatment

SUMMARY:
During 3D-conformal external beam radiation therapy treatments for prostate cancer, the prostate gland moves. The purpose of this study is to determine whether the placement of a prostate immobilization device into the rectum during radiation treatments will decrease the risk of rectal bleeding that is sometimes seen as a late effect from radiation.

DETAILED DESCRIPTION:
* MRI using an endorectal coil done prior to treatment for staging.
* Baseline Quality of Life (QOL) assessment will be completed prior to treatment.
* Total androgen suppression is initiated and will continue for at least 6 months.
* Prostate Immobilization Device (PID) placed during the planning session.
* PID will be placed daily for the first 15 3D external beam radiation treatments.
* QOL assessment and follow-up will take place every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer
* Clinical Stage T1 - T4
* Negative bone scan
* PSA and routine blood work
* >30 years of age
* ECOG Performance 0,1, or 2
* No prior pelvic radiation
* No pacemaker

Exclusion Criteria:

* Inflammatory bowel disease (Crohns, or Ulcerative Colitis)
* Prostatic rectal fistula
* Stricture of anal canal

Ages: 31 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-04; Primary Completion 2005-01 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Rectal toxicity at six month intervals | 2 years

SECONDARY OUTCOMES:
Quality of Life | 2 years
urinary symptoms | 2 years
sexual dysfunction at six month intervals | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V. D'Amico, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute

REFERENCES:
- [Background] Woel R, Beard C, Chen MH, Hurwitz M, Loffredo M, McMahon E, Ching J, Lopes L, D'Amico AV. Acute gastrointestinal, genitourinary, and dermatological toxicity during dose-escalated 3D-conformal radiation therapy (3DCRT) using an intrarectal balloon for prostate gland localization and immobilization. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):392-6. doi: 10.1016/j.ijrobp.2004.10.003. PMID 15890580